CLINICAL TRIAL: NCT00882908
Title: A Phase IIb, Randomized, Double-Blind, Placebo-Controlled Trial to Investigate the Efficacy, Tolerability, Safety and Pharmacokinetics of TMC435 as Part of a Treatment Regimen Including Peginterferon Alfa-2a and Ribavirin In Treatment-Naive Genotype 1 Hepatitis C-Infected Subjects
Brief Title: A Study of TMC435 in Combination With Pegylated Interferon Alp\Fa-2a and Ribavirin in Patients Infected With Genotype 1 Hepatitis C Virus Who Never Received Treatment
Acronym: PILLAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR015799; TMC435-TiDP16-C205 (Other: Tibotec Pharmaceuticals, Ireland); 2008-007147-13 (EudraCT Number)
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Results first posted 2014-06-16 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-05

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; TMC435; Peginterferon alpha-2a; PegIFNalpha-2a; RBV; Ribavirin; Placebo
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir; Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- TMC435 75 mg 12 Wks + PR 24/48 (Experimental): Participants will receive TMC435 75 mg once daily with PegIFNα-2a (P) once weekly and ribavirin (R) twice daily for 12 weeks followed by Placebo once daily and PR for 12 weeks. Treatment with PR was stopped at Week 24 for participants who met response-guided treatment (RGT) criteria. All other participants continued PR until Week 48.
  Interventions: Drug: TMC435; Drug: Ribavirin (R); Drug: PegIFNα-2a (P); Drug: Placebo
- TMC435 75 mg 24 Wks + PR 24/48 (Experimental): Participants will receive TMC435 75 mg once daily with PegIFNα-2a (P) once weekly and ribavirin (R) twice daily for 24 weeks. Treatment with PR was stopped at Week 24 for participants who met response-guided treatment (RGT) criteria. All other participants continued PR until Week 48.
  Interventions: Drug: TMC435; Drug: Ribavirin (R); Drug: PegIFNα-2a (P); Drug: Placebo
- TMC435 150 mg 12 Wks + PR 24/48 (Experimental): Participants will receive TMC435 150 mg once daily with PegIFNα-2a (P) once weekly and ribavirin (R) twice daily for 12 weeks followed Placebo and PR for 12 weeks. Treatment with PR was stopped at Week 24 for participants who met response-guided treatment (RGT) criteria. All other participants continued PR until Week 48.
  Interventions: Drug: TMC435; Drug: Ribavirin (R); Drug: PegIFNα-2a (P); Drug: Placebo
- TMC435 150 mg 24 Wks + PR 24/48 (Experimental): Participants will receive TMC435 150 mg once daily with PegIFNα-2a (P) and ribavirin (R) for 24 weeks. Treatment with PR was stopped at Week 24 for participants who met response-guided treatment (RGT) criteria. All other participants continued PR until Week 48.
  Interventions: Drug: TMC435; Drug: Ribavirin (R); Drug: PegIFNα-2a (P); Drug: Placebo
- Placebo 24 Wks + PR48 (Placebo Comparator): Participants will receive Placebo once daily with PegIFNα-2a (P) and ribavirin (R) for 24 weeks followed by PR until Week 48.
  Interventions: Drug: Ribavirin (R); Drug: PegIFNα-2a (P); Drug: Placebo

INTERVENTIONS:
Drug: TMC435 — TMC435 will be administered as one or two 75 mg capsules orally, once daily, for 12 or 24 weeks.
  Other Names: TMC 435
  Arms: TMC435 150 mg 12 Wks + PR 24/48; TMC435 150 mg 24 Wks + PR 24/48; TMC435 75 mg 12 Wks + PR 24/48; TMC435 75 mg 24 Wks + PR 24/48
Drug: Ribavirin (R) — Ribavirin (R) will be administered as 200 mg tablets (5 to 6 tablets) orally, twice daily, for 48 weeks.
  Other Names: COPEGUS
Drug: PegIFNα-2a (P) — PegIFNα-2a (P) 180 micrograms will be administered as a subcutaneous (under the skin) injection, once weekly for 48 weeks.
  Other Names: PEGASYS
Drug: Placebo — Placebo capsules identical in appearance to TMC435 capsule will be administered orally, once daily, for 48 weeks.

SUMMARY:
The purpose of this study is to evaluate the efficacy of 4 different regimens of TMC435 in combination with peginterferon alfa-2a (PegIFNα-2a) and ribavirin (RBV), defined as the proportion of patients with sustained virologic response at Week 72 (patients with undetectable plasma HCV RNA [less than 25 IU per mL undetectable] at the end of treatment and at Week 72), compared to the control group receiving PegIFN and RBV in combination with TMC435-matched placebo.

DETAILED DESCRIPTION:
This is a randomized (study medication assigned by chance), 5-arm, double-blind (neither investigator nor the participant knows the treatment that the participant receives), placebo-controlled (an inactive substance that is compared with the study medication to test whether the study medication has a real effect in clinical study) study to compare the efficacy, tolerability and safety of different TMC435 regimens combined with peginterferon alfa-2a (PegIFNα-2a) and ribavirin (RBV) versus PegIFNα-2a plus RBV alone in adult treatment-naive patients with chronic genotype 1 HCV infection. The study mainly consists of 3 phases: screening phase (approximately 6 weeks), treatment phase (up to 48 weeks), and follow up phase (up to 48 weeks). In the treatment phase, patients will be divided in to 5 different arms in a 1:1:1:1:1 randomized ratio. In treatment arms 1 and 2, patients will receive 12 weeks of therapy with TMC435 along with PegIFNα 2a and RBV followed by treatment with PegIFNα 2a, RBV, and TMC435-matched placebo. In treatment arms 3 and 4, patients will receive 24 weeks of therapy with TMC435, PegIFNα 2a, and RBV. In treatment arm 5 (control group), patients will receive PegIFNα 2a and RBV for 48 weeks and TMC435 matched placebo for the first 24 weeks. Collection of blood samples for efficacy evaluations will be done at scheduled visits throughout the study. Safety evaluations for adverse events, clinical laboratory tests, physical examination, vital signs and electrocardiogram will be monitored throughout the study. The total duration of the study will be up to approximately 72 weeks after initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented chronic genotype-1 hepatitis C infection and with plasma HCV RNA of > 100,000 IU/mL at screening
* Patients that have not been treated before for HCV
* Patients that are of childbearing potential or have a partner of childbearing potential should agree to use 2 effective methods of contraception

Exclusion Criteria:

* Patients with cirrhosis or evidence of hepatic decompensation
* Co-infection with the human immunodeficiency virus (HIV)
* Any contraindication to Pegasys or Copegus therapy
* History of, or any current medical condition which could impact the safety of the patient in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals, Ireland Clinical Trial, Study Director — Tibotec Pharmaceuticals, Ireland
Locations (71):
- United States (12):
  - Los Angeles, California
  - Jacksonville, Florida
  - Orlando, Florida
  - Palm Harbor, Florida
  - Chicago, Illinois
  - New Orleans, Louisiana
  - Saint Paul, Minnesota
  - New York, New York
  - Chapel Hill, North Carolina
  - Cincinnati, Ohio
  - Germantown, Tennessee
  - Charlottesville, Virginia
- Australia (6):
  - Concord
  - Darlinghurst
  - Fitzroy
  - Melbourne
  - Sydney
  - Woolloongabba
- Vienna, Austria
- Belgium (6):
  - Bruges
  - Brussels
  - Edegem
  - Ghent
  - Leuven
  - Roeselare
- Canada (3):
  - Calgary, Alberta
  - Toronto, Ontario
  - Montreal, Quebec
- Denmark (5):
  - Aarhus
  - Copenhagen
  - Hvidovre
  - Kolding
  - Odense
- France (7):
  - Clichy
  - Créteil
  - Grenoble
  - Lyon
  - Nice
  - Paris
  - Vandœuvre-lès-Nancy
- Germany (9):
  - Berlin
  - Cologne
  - Düsseldorf
  - Frankfurt A. M.
  - Freiburg im Breisgau
  - Hamburg
  - Hanover
  - Stuttgart
  - Würzburg
- New Zealand (3):
  - Auckland
  - Christchurch
  - Hamilton
- Norway (4):
  - Bergen
  - Nordbyhagen
  - Oslo
  - Tromsø
- Poland (6):
  - Bialystok
  - Bydgoszcz
  - Czeladź
  - Kielce
  - Lodz
  - Warsaw
- Russia (5):
  - Moscow
  - Nizhny Novgorod
  - Saint Petersburg
  - Samara
  - Smolensk
- Spain (4):
  - Barcelona
  - Madrid
  - Seville
  - Valencia

REFERENCES:
- [Derived] Lenz O, Verbinnen T, Fevery B, Tambuyzer L, Vijgen L, Peeters M, Buelens A, Ceulemans H, Beumont M, Picchio G, De Meyer S. Virology analyses of HCV isolates from genotype 1-infected patients treated with simeprevir plus peginterferon/ribavirin in Phase IIb/III studies. J Hepatol. 2015 May;62(5):1008-14. doi: 10.1016/j.jhep.2014.11.032. Epub 2014 Nov 28. PMID 25445400
- [Derived] Scott J, Rosa K, Fu M, Cerri K, Peeters M, Beumont M, Zeuzem S, Evon DM, Gilles L. Fatigue during treatment for hepatitis C virus: results of self-reported fatigue severity in two Phase IIb studies of simeprevir treatment in patients with hepatitis C virus genotype 1 infection. BMC Infect Dis. 2014 Aug 26;14:465. doi: 10.1186/1471-2334-14-465. PMID 25164700
- [Derived] Fried MW, Buti M, Dore GJ, Flisiak R, Ferenci P, Jacobson I, Marcellin P, Manns M, Nikitin I, Poordad F, Sherman M, Zeuzem S, Scott J, Gilles L, Lenz O, Peeters M, Sekar V, De Smedt G, Beumont-Mauviel M. Once-daily simeprevir (TMC435) with pegylated interferon and ribavirin in treatment-naive genotype 1 hepatitis C: the randomized PILLAR study. Hepatology. 2013 Dec;58(6):1918-29. doi: 10.1002/hep.26641. Epub 2013 Oct 11. PMID 23907700

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 79 sites in 13 countries: Australia, New Zealand, Canada, Austria, Belgium, Germany, Spain, France, Poland, Russia, Norway, Denmark, and the United States. Approximately 68% of participants were enrolled in Europe, 21% in North America, and 11% in Australia/New Zealand.
Pre-assignment Details: In total, 506 participants were screened; 388 participants were randomized of whom 386 participants started treatment. Two randomized participants did not start treatment due to withdrawal of consent.
Groups:
- TMC435 75 mg 12 Wks + PR 24/48: Participants received TMC435 75 mg once daily with PegIFNα-2a (P) once weekly and ribavirin (R) twice daily for 12 weeks followed by Placebo once daily and PR for 12 weeks. Treatment with PR was stopped at Week 24 for participants who met response-guided treatment (RGT) criteria. All other participants continued PR until Week 48.
- TMC435 75 mg 24 Wks + PR 24/48: Participants received TMC435 75 mg once daily with PegIFNα-2a (P) once weekly and ribavirin (R) twice daily for 24 weeks. Treatment with PR was stopped at Week 24 for participants who met response-guided treatment (RGT) criteria. All other participants continued PR until Week 48.
- TMC435 150 mg 12 Wks + PR 24/48: Participants received TMC435 150 mg once daily with PegIFNα-2a (P) once weekly and ribavirin (R) twice daily for 12 weeks followed Placebo and PR for 12 weeks. Treatment with PR was stopped at Week 24 for participants who met response-guided treatment (RGT) criteria. All other participants continued PR until Week 48.
- TMC435 150 mg 24 Wks + PR 24/48: Participants received TMC435 150 mg once daily with PegIFNα-2a (P) and ribavirin (R) for 24 weeks. Treatment with PR was stopped at Week 24 for participants who met response-guided treatment (RGT) criteria. All other participants continued PR until Week 48.
- Placebo 24 Wks + PR48: Participants received Placebo once daily with PegIFNα-2a (P) and ribavirin (R) for 24 weeks followed by PR until Week 48.
Period: Overall Study
Arm/Group | TMC435 75 mg 12 Wks + PR 24/48 | TMC435 75 mg 24 Wks + PR 24/48 | TMC435 150 mg 12 Wks + PR 24/48 | TMC435 150 mg 24 Wks + PR 24/48 | Placebo 24 Wks + PR48
Started | 78 | 75 | 77 | 79 | 77
Completed | 75 | 69 | 70 | 72 | 71
Not Completed | 3 | 6 | 7 | 7 | 6
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 3 | 5 | 3 | 1 | 2
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 5 | 2
Not completed — Subject reached a virologic endpoint | 0 | 0 | 0 | 0 | 1
Not completed — Study terminated in error | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TMC435 75 mg 12 Wks + PR 24/48 | TMC435 75 mg 24 Wks + PR 24/48 | TMC435 150 mg 12 Wks + PR 24/48 | TMC435 150 mg 24 Wks + PR 24/48 | Placebo 24 Wks + PR48 | Total
Number analyzed (Participants) | 78 | 75 | 77 | 79 | 77 | 386
Age, Continuous [Median (Full Range); unit: years] | 47 [19 to 66] | 46 [18 to 67] | 47 [18 to 69] | 47 [18 to 69] | 45 [21 to 67] | 46.5 [18 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 28 | 34 | 35 | 38 | 173
  Male | 40 | 47 | 43 | 44 | 39 | 213
Region of Enrollment [Number; unit: participants]
  Asia Pacific | 9 | 9 | 7 | 13 | 4 | 42
  Europe | 52 | 52 | 56 | 44 | 58 | 262
  North-America | 17 | 14 | 14 | 22 | 15 | 82

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Achieving a Sustained Virologic Response at Week 72 (SVRW72)
Description: The table below shows the percentage of participants in each treatment group who achieved a SVRW72, defined as the percentage of participants with undetectable plasma Hepatitis C virus ribonucleic acid levels at end of treatment (EOT) and at Week 72.
Time Frame: Week 72
Population: The intent-to treat population (defined as those participants who received at least 1 dose of study medication) was used for all efficacy and safety analyses.
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 75 mg 12 Wks + PR 24/48 | TMC435 75 mg 24 Wks + PR 24/48 | TMC435 150 mg 12 Wks + PR 24/48 | TMC435 150 mg 24 Wks + PR 24/48 | Placebo 24 Wks + PR48
Number analyzed (Participants) | 78 | 75 | 77 | 79 | 77
Percentage of participants | 80.8 | 70.7 | 77.9 | 84.8 | 64.9
Statistical Analysis 1: Comparison: TMC435 75 mg 12 Wks + PR 24/48 vs TMC435 75 mg 24 Wks + PR 24/48 vs Placebo 24 Wks + PR48; TMC435 75 mg 12 and 24 week treatment groups were pooled and the percentage of participants acheiving SVRW72 were compared with the percentage of participants acheiving SVRW72 in the placebo treatment group; Test type: Superiority or Other; p = 0.051, Regression, Logistic; Difference in proportions of SVRW72 = 13.0, 97.5% CI 2-sided [-1.9 to 28.0] — Difference in percentages of participants in the TMC435 75mg and placebo groups with undetectable plasma Hepatitis C virus ribonucleic acid levels at end of treatment (EOT) and at Week 72 estimated from the logistic regression model
Statistical Analysis 2: Comparison: TMC435 150 mg 12 Wks + PR 24/48 vs TMC435 150 mg 24 Wks + PR 24/48 vs Placebo 24 Wks + PR48; TMC/PR 150 mg 12 and 24 week treatment groups were pooled and the percentage of participants achieving SVRW72 was compared the percentage of participants achieving SVRW72 in the placebo treatment group; Test type: Superiority or Other; p = 0.004, Regression, Logistic; Difference in proportions of SVRW72 = 18.9, 97.5% CI 2-sided [4.4 to 33.5] — Difference in percentages of participants in the TMC435 150mg and placebo groups with undetectable plasma Hepatitis C virus ribonucleic acid levels at end of treatment (EOT) and at Week 72 estimated from the logistic regression model

2. Secondary Outcome: The Percentage of Participants Achieving Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels of Less Than 25 IU/mL Undetectable During Treatment and Follow-up
Description: The table below shows the percentage of participants in each treatment group who achieved plasma HCV RNA levels of less than 25 IU/mL undetectable at selected time points during treatment, follow-up, and at end of treatment (EOT).
Time Frame: Weeks, 2, 4, 8, 12, 24, 36, 48, 60, 72, and at EOT (up to Week 24 or 48)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 75 mg 12 Wks + PR 24/48 | TMC435 75 mg 24 Wks + PR 24/48 | TMC435 150 mg 12 Wks + PR 24/48 | TMC435 150 mg 24 Wks + PR 24/48 | Placebo 24 Wks + PR48
Number analyzed (Participants) | 78 | 75 | 77 | 79 | 77
Percentage of participants
  Week 2 | 39.7 | 30.7 | 23.4 | 39.2 | 2.6
  Week 4 | 75.6 | 68.0 | 75.3 | 74.7 | 5.2
  Week 8 | 87.2 | 90.7 | 92.2 | 93.7 | 26.0
  Week 12 | 91.0 | 93.3 | 93.5 | 94.9 | 55.8
  Week 24 | 92.3 | 93.3 | 84.4 | 87.3 | 77.9
  Week 36 | 85.9 | 81.3 | 81.8 | 84.8 | 76.6
  Week 48 | 79.5 | 77.3 | 79.2 | 82.3 | 74.0
  Week 60 | 79.5 | 68.0 | 75.3 | 83.5 | 63.6
  Week 72 | 79.5 | 70.7 | 77.9 | 82.3 | 64.9
  EOT (up to Week 24 or 48) | 92.3 | 97.3 | 92.2 | 93.7 | 79.2

3. Secondary Outcome: The Percentage of Participants Who Achieved Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels of Less Than 25 IU/mL Detectable or Undetectable During Treatment and Follow-up
Description: The table below shows the percentage of participants in each treatment group who achieved plasma levels of HCV RNA less than 25 IU/mL detectable or undetectable at selected time points during treatment, follow-up, and at end of treatment (EOT).
Time Frame: Weeks 2, 4, 8, 12, 24, 36, 48, 60, 72, and at EOT (up to Week 24 or 48)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 75 mg 12 Wks + PR 24/48 | TMC435 75 mg 24 Wks + PR 24/48 | TMC435 150 mg 12 Wks + PR 24/48 | TMC435 150 mg 24 Wks + PR 24/48 | Placebo 24 Wks + PR48
Number analyzed (Participants) | 78 | 75 | 77 | 79 | 77
Percentage of participants
  Week 2 | 65.4 | 66.7 | 75.3 | 78.5 | 5.2
  Week 4 | 85.9 | 88.0 | 90.9 | 91.1 | 15.6
  Week 8 | 93.6 | 94.7 | 93.5 | 93.7 | 49.4
  Week 12 | 93.6 | 94.7 | 96.1 | 94.9 | 66.2
  Week 24 | 92.3 | 93.3 | 84.4 | 89.9 | 80.5
  Week 36 | 85.9 | 81.3 | 81.8 | 84.8 | 79.2
  Week 48 | 79.5 | 77.3 | 79.2 | 82.3 | 75.3
  Week 60 | 79.5 | 68.0 | 75.3 | 83.5 | 64.9
  Week 72 | 79.5 | 70.7 | 77.9 | 83.5 | 64.9
  EOT (up to Week 24 or 48) | 93.6 | 97.3 | 92.2 | 96.2 | 83.1

4. Secondary Outcome: The Percentage of Participants Achieving Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels of Greater Than or Equal to 2 log10 Drop During Treatment
Description: The table below shows the percentage of participants in each treatment group who achieved plasma levels of HCV RNA greater than or equal to 2 log10 drop from Baseline at selected time points during treatment.
Time Frame: Baseline (Day 1) and Weeks, 2, 4, 8, and 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 75 mg 12 Wks + PR 24/48 | TMC435 75 mg 24 Wks + PR 24/48 | TMC435 150 mg 12 Wks + PR 24/48 | TMC435 150 mg 24 Wks + PR 24/48 | Placebo 24 Wks + PR48
Number analyzed (Participants) | 78 | 75 | 77 | 79 | 77
Percentage of participants
  Week 2 | 93.6 | 98.7 | 97.4 | 98.7 | 40.3
  Week 4 | 94.9 | 98.7 | 97.4 | 93.7 | 71.4
  Week 8 | 97.4 | 97.3 | 97.4 | 94.9 | 84.4
  Week 12 | 97.4 | 96.0 | 96.1 | 96.2 | 89.6

5. Secondary Outcome: The Percentage of Participants Who Achieved a Sustained Virologic Response 24 Weeks After the Planned End of Treatment (SVR24)
Description: The table below shows the percentage of participants in each treatment group who achieved a SVR24, defined as having undetectable plasma Hepatitis C virus ribonucleic acid levels at the end of treatment (EOT) and 24 weeks after the EOT.
Time Frame: Week 48 or 72
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 75 mg 12 Wks + PR 24/48 | TMC435 75 mg 24 Wks + PR 24/48 | TMC435 150 mg 12 Wks + PR 24/48 | TMC435 150 mg 24 Wks + PR 24/48 | Placebo 24 Wks + PR48
Number analyzed (Participants) | 78 | 75 | 77 | 79 | 77
Percentage of participants | 82.1 | 74.7 | 80.5 | 86.1 | 64.9

6. Secondary Outcome: The Percentage of Participants Achieving a Rapid Virologic Response (RVR)
Description: The table below shows the percentage of participants in each treatment group who achieved a RVR, defined as having undetectable plasma Hepatitis C virus ribonucleic acid levels after receiving 4 weeks of treatment.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 75 mg 12 Wks + PR 24/48 | TMC435 75 mg 24 Wks + PR 24/48 | TMC435 150 mg 12 Wks + PR 24/48 | TMC435 150 mg 24 Wks + PR 24/48 | Placebo 24 Wks + PR48
Number analyzed (Participants) | 78 | 75 | 77 | 79 | 77
Percentage of participants | 75.6 | 68.0 | 75.3 | 74.7 | 5.2

7. Secondary Outcome: The Percentage of Participants Achieving an Early Virologic Response (EVR)
Description: The table below shows the percentage of participants who achieved an EVR, defined as having a change from baseline in plasma Hepatitis C virus ribonucleic acid of 2 log10 at Week 12.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 75 mg 12 Wks + PR 24/48 | TMC435 75 mg 24 Wks + PR 24/48 | TMC435 150 mg 12 Wks + PR 24/48 | TMC435 150 mg 24 Wks + PR 24/48 | Placebo 24 Wks + PR48
Number analyzed (Participants) | 78 | 75 | 77 | 79 | 77
Percentage of participants | 97.4 | 96.0 | 96.1 | 96.2 | 89.6

8. Secondary Outcome: The Percentage of Participants Achieving a Complete Early Virologic Response (cEVR)
Description: The table below shows the percentage of participants in each treatment group who had a cEVR, defined as having undetectable plasma Hepatitis C Virus ribonucleic acid levels at Week 12.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 75 mg 12 Wks + PR 24/48 | TMC435 75 mg 24 Wks + PR 24/48 | TMC435 150 mg 12 Wks + PR 24/48 | TMC435 150 mg 24 Wks + PR 24/48 | Placebo 24 Wks + PR48
Number analyzed (Participants) | 78 | 75 | 77 | 79 | 77
Percentage of participants | 91.0 | 93.3 | 93.5 | 94.9 | 55.8

9. Secondary Outcome: The Percentage of Participants Achieving a Sustained Virologic Response 12 Weeks After the Planned End of Treatment (SVR12)
Description: The table below shows the percentage of participants who achieved undetectable plasma Hepatitis C virus ribonucleic acid levels at the end of treatment (EOT) and 12 Weeks after the EOT.
Time Frame: Up to Week 36 or 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 75 mg 12 Wks + PR 24/48 | TMC435 75 mg 24 Wks + PR 24/48 | TMC435 150 mg 12 Wks + PR 24/48 | TMC435 150 mg 24 Wks + PR 24/48 | Placebo 24 Wks + PR48
Number analyzed (Participants) | 78 | 75 | 77 | 79 | 77
Percentage of participants | 83.3 | 76.0 | 80.5 | 86.1 | 66.2

10. Secondary Outcome: Number of Participants With Viral Breakthrough
Description: The table below shows the number of participants in each treatment group who experienced viral breakthrough during the TMC435 treatment period of the study, defined as a confirmed increase of more than 1 log10 IU/mL in plasma Hepatitis C virus (HCV) ribonucleic acid (RNA) level from the lowest level reached or a confirmed value of plasma HCV RNA more than 100 IU/mL in participants whose plasma HCV RNA level had previously been below the limit of quantification (less than 25 IU/mL detectable or undetectable).
Time Frame: Week 24 or 48
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | TMC435 75 mg 12 Wks + PR 24/48 | TMC435 75 mg 24 Wks + PR 24/48 | TMC435 150 mg 12 Wks + PR 24/48 | TMC435 150 mg 24 Wks + PR 24/48 | Placebo 24 Wks + PR48
Number analyzed (Participants) | 78 | 75 | 77 | 79 | 77
Participants | 5 | 2 | 6 | 2 | 4

11. Secondary Outcome: The Number of Participants With Viral Relapse
Description: The table below shows the number of participants who experienced viral relapse, defined as a confirmed detectable plasma Hepatitis C virus (HCV) ribonucleic acid (RNA) level during the follow-up period in participants with undetectable plasma HCV RNA (less than 25 IU/mL undetectable) at the end of treatment.
Time Frame: Up to Week 72
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | TMC435 75 mg 12 Wks + PR 24/48 | TMC435 75 mg 24 Wks + PR 24/48 | TMC435 150 mg 12 Wks + PR 24/48 | TMC435 150 mg 24 Wks + PR 24/48 | Placebo 24 Wks + PR48
Number analyzed (Participants) | 78 | 75 | 77 | 79 | 77
Participants | 8 | 14 | 6 | 6 | 11

12. Secondary Outcome: The Number of Participants With Abnormal Alanine Aminotransferase (ALT) Levels at Baseline Who Achieved Normalized ALT Levels at the End of Treatment (EOT)
Description: The table below shows the number of participants with abnormal ALT levels at Baseline who achieved ALT levels within the normal range at the EOT.
Time Frame: Baseline (Day 1) up to Week 24 or 48
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- All TMC435 Treatment Groups: Participants in all 4 TMC435 treatment groups combined.
Arm/Group | TMC435 75 mg 12 Wks + PR 24/48 | TMC435 75 mg 24 Wks + PR 24/48 | TMC435 150 mg 12 Wks + PR 24/48 | TMC435 150 mg 24 Wks + PR 24/48 | All TMC435 Treatment Groups
Number analyzed (Participants) | 43 | 45 | 48 | 43 | 179
Participants | 39 | 37 | 39 | 35 | 150

13. Secondary Outcome: Plasma Concentrations of TMC435
Description: The table below shows median (range) predose plasma concentration (C0h) values and median (range) average steady-state plasma concentration (Css,av) values for participants in each of the 4 TMC435 treatment groups.
Time Frame: Two random blood samples taken at least 2 hours apart at Weeks 2, 4, 8, 12, 16, and 24
Population: Participants who received at least 1 dose of study medication with at least 1 post-baseline pharmacokinetic (PK) assessment were included in the PK analysis population.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | TMC435 75 mg 12 Wks + PR 24/48 | TMC435 75 mg 24 Wks + PR 24/48 | TMC435 150 mg 12 Wks + PR 24/48 | TMC435 150 mg 24 Wks + PR 24/48
Number analyzed (Participants) | 77 | 75 | 77 | 78
ng/mL
  Coh | 240.9 [0 to 1927] | 213.6 [40 to 2124] | 1123.3 [91 to 13771] | 1176.7 [0 to 9875]
  Css, av | 413.6 [6 to 2091] | 374.0 [151 to 2385] | 1661.8 [123 to 15868] | 1501.6 [47 to 11648]

14. Secondary Outcome: Area Under the Plasma Concentration-time Curve From 0 to 24 Hours (AUC24h) for TMC435
Description: The table below shows the median (range) AUC24h values for TMC435 for participants in each of the 4 TMC435 treatment groups. Two blood samples taken at least 2 hours apart from each other for determination of TMC435 plasma pharmacokinetics were obtained in all participants on Weeks 2, 4, 8, 12, 16, and 24 to obtain Bayesian estimates of TMC435 AUC24h (overall exposure).
Time Frame: Two random blood samples taken at least 2 hours apart at Weeks 2, 4, 8, 12, 16, and 24
Population: as for outcome 13
Measure: Median (Full Range); unit: ng*h/mL
Arm/Group | TMC435 75 mg 12 Wks + PR 24/48 | TMC435 75 mg 24 Wks + PR 24/48 | TMC435 150 mg 12 Wks + PR 24/48 | TMC435 150 mg 24 Wks + PR 24/48
Number analyzed (Participants) | 77 | 75 | 77 | 78
ng*h/mL | 9926.4 [138 to 50179] | 8976.8 [3615 to 57243] | 39884.0 [2948 to 380830] | 36038.8 [1134 to 279550]

ADVERSE EVENTS:
Time Frame: 72 weeks
Description: All participants who received at least one dose of investigational medication included in safety analysis.
Arm/Group | TMC435 75 mg 12 Wks + PR 24/48 | TMC435 75 mg 24 Wks + PR 24/48 | TMC435 150 mg 12 Wks + PR 24/48 | TMC435 150 mg 24 Wks + PR 24/48 | Placebo 24 Wks + PR48
Serious Adverse Events (participants affected / at risk) | 9/78 | 4/75 | 4/77 | 3/79 | 10/77
Other Adverse Events (participants affected / at risk) | 76/78 | 75/75 | 74/77 | 77/79 | 75/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TMC435 75 mg 12 Wks + PR 24/48 (N=78) | TMC435 75 mg 24 Wks + PR 24/48 (N=75) | TMC435 150 mg 12 Wks + PR 24/48 (N=77) | TMC435 150 mg 24 Wks + PR 24/48 (N=79) | Placebo 24 Wks + PR48 (N=77)
Incision site cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Perihepatic abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Vulval abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Ocular vasculitis (Eye disorders) | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Myopericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TMC435 75 mg 12 Wks + PR 24/48 (N=78) | TMC435 75 mg 24 Wks + PR 24/48 (N=75) | TMC435 150 mg 12 Wks + PR 24/48 (N=77) | TMC435 150 mg 24 Wks + PR 24/48 (N=79) | Placebo 24 Wks + PR48 (N=77)
Fatigue (General disorders) | 26 | 35 | 32 | 38 | 37
Influenza like illness (General disorders) | 21 | 32 | 18 | 27 | 29
Pyrexia (General disorders) | 18 | 15 | 15 | 16 | 13
Asthenia (General disorders) | 20 | 12 | 18 | 13 | 16
Irritability (General disorders) | 10 | 7 | 14 | 11 | 8
Chills (General disorders) | 4 | 8 | 6 | 7 | 8
Injection site erythema (General disorders) | 4 | 8 | 5 | 7 | 4
Injection site reaction (General disorders) | 5 | 4 | 2 | 2 | 4
Pain (General disorders) | 6 | 2 | 2 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 25 | 17 | 30 | 24 | 35
Rash (Skin and subcutaneous tissue disorders) | 21 | 10 | 16 | 18 | 18
Dry skin (Skin and subcutaneous tissue disorders) | 12 | 12 | 17 | 22 | 14
Alopecia (Skin and subcutaneous tissue disorders) | 20 | 11 | 11 | 11 | 16
Erythema (Skin and subcutaneous tissue disorders) | 3 | 2 | 5 | 5 | 4
Eczema (Skin and subcutaneous tissue disorders) | 7 | 1 | 3 | 3 | 5
Pruritus generalised (Skin and subcutaneous tissue disorders) | 3 | 2 | 3 | 6 | 5
Night sweats (Skin and subcutaneous tissue disorders) | 6 | 1 | 1 | 2 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 4 | 1 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 3 | 4
Headache (Nervous system disorders) | 41 | 34 | 35 | 32 | 40
Dizziness (Nervous system disorders) | 10 | 3 | 4 | 12 | 6
Disturbance in attention (Nervous system disorders) | 5 | 3 | 6 | 4 | 3
Dysgeusia (Nervous system disorders) | 6 | 1 | 5 | 4 | 5
Paraesthesia (Nervous system disorders) | 1 | 0 | 4 | 1 | 1
Syncope (Nervous system disorders) | 1 | 2 | 2 | 1 | 4
Migraine (Nervous system disorders) | 0 | 0 | 1 | 4 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 4
Nausea (Gastrointestinal disorders) | 26 | 16 | 20 | 24 | 21
Diarrhoea (Gastrointestinal disorders) | 12 | 14 | 11 | 10 | 12
Vomiting (Gastrointestinal disorders) | 5 | 3 | 6 | 8 | 5
Dry mouth (Gastrointestinal disorders) | 5 | 7 | 3 | 6 | 7
Abdominal pain upper (Gastrointestinal disorders) | 5 | 4 | 6 | 4 | 4
Dyspepsia (Gastrointestinal disorders) | 4 | 5 | 4 | 6 | 6
Constipation (Gastrointestinal disorders) | 6 | 1 | 7 | 2 | 5
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 4 | 3 | 4
Aphthous stomatitis (Gastrointestinal disorders) | 2 | 1 | 4 | 2 | 3
Insomnia (Psychiatric disorders) | 19 | 14 | 23 | 13 | 23
Depression (Psychiatric disorders) | 8 | 4 | 9 | 11 | 14
Sleep disorder (Psychiatric disorders) | 8 | 3 | 4 | 7 | 4
Mood altered (Psychiatric disorders) | 4 | 5 | 1 | 8 | 7
Depressed mood (Psychiatric disorders) | 4 | 4 | 3 | 6 | 3
Anxiety (Psychiatric disorders) | 5 | 2 | 4 | 4 | 5
Mood swings (Psychiatric disorders) | 4 | 0 | 1 | 5 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 17 | 12 | 16 | 10 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 12 | 14 | 16 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 8 | 10 | 7 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1 | 4 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 3 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 3 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 9 | 12 | 13 | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 8 | 7 | 6 | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 | 9 | 10 | 5 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 4 | 4 | 8
Neutropenia (Blood and lymphatic system disorders) | 15 | 23 | 19 | 18 | 16
Anaemia (Blood and lymphatic system disorders) | 15 | 16 | 17 | 15 | 16
Leukopenia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 6 | 4
Nasopharyngitis (Infections and infestations) | 1 | 5 | 4 | 4 | 6
Influenza (Infections and infestations) | 1 | 5 | 4 | 3 | 3
Urinary tract infection (Infections and infestations) | 2 | 2 | 1 | 5 | 2
Sinusitis (Infections and infestations) | 4 | 0 | 1 | 2 | 2
Weight decreased (Investigations) | 7 | 3 | 3 | 6 | 3
Neutrophil count decreased (Investigations) | 1 | 5 | 5 | 4 | 4
Blood bilirubin increased (Investigations) | 1 | 0 | 5 | 5 | 0
Alanine aminotransferase increased (Investigations) | 3 | 1 | 1 | 5 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 1 | 6 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 4 | 0
Anorexia (Metabolism and nutrition disorders) | 10 | 12 | 11 | 9 | 11
Decreased appetite (Metabolism and nutrition disorders) | 6 | 3 | 4 | 4 | 6
Dry eye (Eye disorders) | 3 | 2 | 3 | 4 | 4
Vision blurred (Eye disorders) | 3 | 1 | 5 | 3 | 1
Vertigo (Ear and labyrinth disorders) | 5 | 1 | 3 | 4 | 4
Hot flush (Vascular disorders) | 1 | 0 | 2 | 5 | 2
Hypertension (Vascular disorders) | 0 | 1 | 1 | 4 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0 | 5 | 2 | 2
Hypothyroidism (Endocrine disorders) | 6 | 1 | 1 | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days